CLINICAL TRIAL: NCT02719080
Title: Department of Anesthesiology, Ruijin Hospital, Shanghai JiaoTong University School of Medicine
Brief Title: The Relationship Between Cerebral State and Emotion in Anesthesiologist and Surgeon
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, HoiYin Cheung, doctor, Ruijin Hospital
Other Study IDs: 20160201
Record Dates: First submitted 2016-03-20; First posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Burnout, Professional
Keywords: anaesthetists, surgeons, stress, burnout
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study was designed to observe the cerebral state obtained via wavelet analysis (HXD-I,Beijing Easymonitor Technology Co.Ltd, China) and evaluate the emotion in various states in anesthesiologist and surgeon. And we also explore the association between the characteristic of cerebral state and the emotion.

DETAILED DESCRIPTION:
A total of 20 anesthesiologist (A group) and 20 surgeon(S group) in Ruijin hospital were enrolled for this study. Except had a medical history of mental illness or emotional disorder and pregnant woman. A group and S group completed emotional self-perceived questionnaire and then observe the characteristic of cerebral state via cerebral state monitor. They also completed anonymous questionnaire, including Maslach Burnout Inventory-General Survey(MBI-GS), Self-reporting Inventory-90(SCI-90), Burnout Measure(BM).

ELIGIBILITY:
Inclusion Criteria:

* A total of 20 anesthesiologist (A group) and 20 surgeon(S group) in Ruijin hospital were enrolled for this study.

Exclusion Criteria:

* had a medical history of mental illness or emotional disorder and pregnant woman.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: anesthesiologist and surgeon in Ruijin hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The relationship between cerebral state and emotion in doctors | one week
  subjects completed emotional self-perceived questionnaire and then observe the characteristic of cerebral state via cerebral state monitor. They also completed anonymous questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Luo, M.D.,Ph.D, Study Director — Department of Anesthesiology, Ruijin Hospital, Shanghai JiaoTong University School of Medicine,
Locations (1):
- Department of Anesthesiology, Ruijin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Holmqvist R, Jeanneau M. Burnout and psychiatric staff's feelings towards patients. Psychiatry Res. 2006 Dec 7;145(2-3):207-13. doi: 10.1016/j.psychres.2004.08.012. Epub 2006 Oct 27. PMID 17070932
- [Background] Murray D, Dodds C. The effect of sleep disruption on performance of anaesthetists--a pilot study. Anaesthesia. 2003 Jun;58(6):520-5. doi: 10.1046/j.1365-2044.2003.03131.x. PMID 12846614
- [Background] Mountain SA, Quon BS, Dodek P, Sharpe R, Ayas NT. The impact of housestaff fatigue on occupational and patient safety. Lung. 2007 Jul-Aug;185(4):203-9. doi: 10.1007/s00408-007-9010-5. Epub 2007 May 3. PMID 17476556
- [Background] Candra H, Yuwono M, Handojoseno A, Chai R, Su S, Nguyen HT. Recognizing emotions from EEG subbands using wavelet analysis. Annu Int Conf IEEE Eng Med Biol Soc. 2015;2015:6030-3. doi: 10.1109/EMBC.2015.7319766. PMID 26737666